CLINICAL TRIAL: NCT07009730
Title: Clinical Outcomes Between Pulsatile and Non-Pulsatile Flow During Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Ishwor Thapaliya, Principal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 20.7.2017
Record Dates: First submitted 2025-05-29; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Surgery; Cardiac Surgery Requiring Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiopulmonary bypass, pulsatile flow
  Interventions: Procedure: Bypassing Agents

INTERVENTIONS:
Procedure: Bypassing Agents — Cardiopulmonary bypass surgery, pulsatile flow

SUMMARY:
The aim of this prospective, randomized study was to compare clinical outcomes of Pulsatile and non-pulsatile flow during Cardiopulmonary Bypass.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing Atrial Septal Defect closure and Mitral Valve replacement

Exclusion Criteria:

* • Moderate and severe LVEF
* • Patient with bleeding dysfunction;AKI ;deranged liver dysfunction\
* • Patient/Surrogate decision maker not giving written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients undergoing Atrial Septal Defect closure and mitral Valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
ICU Length of Stay | 12 months
  Measured in days from ICU admission to ICU discharge

SECONDARY OUTCOMES:
Duration of Cardiopulmonary Bypass (CPB) | 12 months
  Measured in minutes from initiation to termination of bypass

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Institute of Medicine (IOM), Kathmandu, Nepal, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Undecided